CLINICAL TRIAL: NCT04761562
Title: Use of Autologous Plasma Rich in Platelets and Extracellular Vesicles in the Surgical Treatment of Chronic Otitis Media
Brief Title: Use of Autologous Plasma Rich in Platelets and Extracellular Vesicles in the Surgical Treatment of Chronic Middle Ear Infections
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana (Other)
Responsible Party: Principal Investigator, Nejc Steiner, Principal Investigator, Resident of otorhinolaryngology, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PVRPTY2021
Record Dates: First submitted 2021-02-12; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Otitis Media Chronic; Tympanic Membrane Perforation
Keywords: Tympanoplasty; Platelet-Rich Plasma
MeSH Terms: conditions — Tympanic Membrane Perforation | interventions — Platelet Count; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Both the patient and the outcomes assessors of the tympanic membrane healing, hearing and questionnaires will not know in which group the patient was placed. The patient group will be known only to the doctoral student, the surgeon and the person who will prepare the PVRP. None of them will be included in the process randomisation and final assessment 3 and 6 months after surgery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Patients will be treated with a standard surgical procedure - tympanoplasty.
  Interventions: Procedure: Control group
- PVRP group (Experimental): Patients will be treated with a standard surgical procedure - tympanoplasty combined with PVRP. PVRP will be applied to the reconstructed tympanic membrane.
  Interventions: Drug: Platelet- and extracellular vesicle-rich plasma

INTERVENTIONS:
Drug: Platelet- and extracellular vesicle-rich plasma — PVRP will initially be applied to the gelatine sponge without prior exogenous activation, which will first be inserted into the middle ear cavity to support the reconstructed tympanic membrane. The remainder of the PVRP will then be exogenously activated with calcium chloride. Gel rich with platelets and extracellular vesicles will be created and applied on top of the reconstructed tympanic membrane. Finally, the external auditory canal will be filled with pieces of gelatine sponge soaked with PVRP.
  Arms: PVRP group
Procedure: Control group — Edges of the tympanic membrane perforation will be refreshed and the tympanomeatal flap raised. Under the tympanic membrane perforation, a guide (fascia of the temporalis muscle, perichondrium, cartilage or fat) will be placed. An absorbent gelatin sponge will be placed under the guide and on the outer surface of the reconstructed tympanic membrane.
  Other Names: Standard tympanoplasty
  Arms: Control group

SUMMARY:
This clinical study evaluates the efficacy of the autologous blood-derived product called platelet- and extracellular vesicle-rich plasma as a supplement to the surgical treatment of chronic tympanic membrane perforations.

Half of the participants will be treated with standard surgical procedure called tympanoplasty and addition of platelet- and extracellular vesicle-rich plasma. Another half will be treated with only the standard tympanoplasty.

DETAILED DESCRIPTION:
The study is designed to be mono-centric, prospective, double-blind, parallel, uniformly randomised, controlled, with a fixed sample.

The purpose of the study is to determine whether autologous platelet- and extracellular vesicle-rich plasma (PVRP) made from peripheral venous blood, promotes healing of tympanic membrane perforations, improves hearing and quality of life after surgical procedure called tympanoplasty.

Tympanoplasty is a surgical procedure in which the surgeon refreshes the edges of the perforation of the eardrum and thus encourage re-healing of the eardrum. The tympanic membrane lies in the air, thus a tissue (muscle fascia, perichondrium, fat or cartilage) has to be put underneath the perforation and eardrum remnant. This then serves as a guide for the newly formed tympanic cells can outgrow the perforation.

Patients attending outpatient examinations will be included in the study if they meet the inclusion criteria. Included patients will be randomised in two groups.

Patients from the control group will be treated with a standard surgical treatment - tympanoplasty. The surgical procedure for the patients from the treatment group will be the same as for the control group, for the exception that PVRP will be added around the tympanic membrane remnant. PVRP will be activated inside (endogenous) and outside (exogenous) the body.

Postoperatively patients will be assessed at examinations using an endoscope, otomicroscope, Chronic otitis media questionnaire and tests of hearing and balance. Laboratory blood tests will determine the presence of possible inflammation and assess the composition of the preparation.

Research hypotheses

* Hypothesis 1: In the group of patients treated with platelet-rich plasma and extracellular vesicles, the proportion of healed tympanic surfaces in terms of initial perforation will be higher than in patients treated without platelet-rich plasma and extracellular vesicles.
* Hypothesis 2: In the group of patients treated with platelet-rich plasma and extracellular vesicles, complete healing of the tympanic membrane will occur to a greater extent than in patients treated without platelet-rich plasma and extracellular vesicles.
* Hypothesis 3: In the group of patients treated with platelet-rich plasma and extracellular vesicles, hearing improvement will be greater than in patients treated with platelet-rich plasma and extracellular vesicles.
* Hypothesis 4: The quality of life of patients with larger perforations assessed with the COMQ-12 questionnaire will be lower than in patients treated without platelet-rich plasma and extracellular vesicles.
* Hypothesis 5: The quality of life assessed by the COMQ-12 questionnaire will be better in the group of patients treated with platelet-rich plasma and extracellular vesicles than in patients treated without platelet-rich plasma and extracellular vesicles.

ELIGIBILITY:
Inclusion Criteria:

* tympanic membrane,
* dry middle ear cavity,
* absence of exclusion criteria.

Exclusion Criteria:

* signs of cholesteatoma,
* anemia,
* thrombocytopenia,
* chronic use of immunomodulatory agents and / or antimicrobials,
* malignancy in the ear area,
* systemic infectious disease,
* autoimmune disease,
* inability and / or refusal of the patient to participate in the research,
* pregnancy and / or breast-feeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-14 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change of tympanic membrane perforation size | Baseline (1 day pre-operatively), 6 weeks, 3 months and 6 months after surgery.
  The size of the tympanic membrane perforation will be expressed as proportion of the total surface area of the tympanic membrane. Number of pixels on an endoscopic photograph of the tympanic membrane will be measured with a computer program. The measured number of perforation pixels will be divided by the measured number of pixels of the entire tympanic membrane. The measurement will be performed by two doctors and the average value of the measured proportion of the drum surface used.
Change in Chronic Otitis Media Questionnaire 12 score | Baseline (1 day pre-operatively), 6 months after surgery.
  * the unabbreviated scale title: Chronic Otitis Media Questionnaire 12
  * the minimum and maximum values: 0, 60
  * higher scores mean a worse outcome.
  Sum score of Chronic Otitis Media Questionnaire 12 (COMQ-12), patient-reported health-related quality of life measure. Questionnaire consists of 12 questions, each question is scored from 0 to 5 points.

SECONDARY OUTCOMES:
Change in hearing threshold level | Baseline (1 day pre-operatively), 6 weeks, 3 months and 6 months after surgery.
  Pure tone audiometry will be done and pure tone average calculated from frequencies 125 to 8000 Herz.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vozel D., Božič D., Jeran M., Jan Z., Pajnič M., Pađen L., Uršič B., Iglič A., Kralj-Iglič V., Battelino S. 2020. Treatment with platelet- and extracellular vesicle-rich plasma in otorhinolaryngology-a review and future perspectives. V Advances in Biomembranes and Lipid Self-Assembly. Academic Press. https://doi.org/10.1016/bs.abl.2020.05.003
- [Background] Vozel D, Steiner N, Bozanic Urbancic N, Mladenov D, Battelino S. Slovenian Cross-Cultural Adaptation and Validation of Health-Related Quality of Life Measures for Chronic Otitis Media (COMQ-12), Vertigo (DHI, NVI) and TINNITUS (THI). Zdr Varst. 2020 Jun 25;59(3):120-127. doi: 10.2478/sjph-2020-0016. eCollection 2020 Sep. PMID 32952712